CLINICAL TRIAL: NCT05783804
Title: Plaque Reversal With Early, Aggressive Lipid Lowering Therapy
Acronym: EAGLE
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, E.S.stroes, Prof. dr. E.S.G. Stroes, MD, PhD., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL75337.018.20
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study evaluates whether plaques in young patients with familial hypercholesterolemia (aged below 50 years) are susceptible to significant plaque regression with early, intensive lipid lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with heterozygous familial hypercholesterolemia
* Adult between 18 and 50 years old
* LDL cholesterol levels above 100 mg/dl (>2.6 mmol/L) at inclusion

Exclusion Criteria:

* Renal insufficiency, defined as eGFR < 30 ml/min
* History of atherosclerotic cardiovascular events
* Atrial fibrillation
* Any other treatment or clinically relevant condition that could interfere with the conduct or interpretation of the study in the opinion of the investigator
* Inability or unwillingness to comply with the protocol requirements, or deemed by investigator to be unfit for the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult (newly diagnosed) heterozygous FH patients between 18 and 50 years with non-calcificated plaque on coronary CT angiography and who are not optimally treated yet.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
CAD Progression | 40 Weeks
  Difference in total plaque volume between the initial and follow-up CCTA scan

SECONDARY OUTCOMES:
Non-calcified plaque progression | 40 Weeks
  Difference in non-calcified plaque volume between the baseline and follow-up CCTA scan
Calcified plaque progression | 40 Weeks
  Difference in calcified plaque volume between the baseline and follow-up CCTA scan
Number of high-risk plaques | 40 Weeks
  Difference in number of high-risk plaques between the baseline and follow-up CCTA scan
Difference in Pericoronary Adipose Tissue Attenuation | 40 Weeks
  Difference in Pericoronary Adipose Tissue Attenuation between the baseline and follow-up CCTA scan

CONTACTS AND LOCATIONS:
Overall Officials: Erik SG Stroes, MD, PhD, Principal Investigator — Amsterdam UMC, location AMC
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands